CLINICAL TRIAL: NCT04660526
Title: RAndomized Cluster Evaluation of Cardiac ARrest Systems
Brief Title: RACE-CARS - RAndomized Cluster Evaluation of Cardiac ARrest Systems
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00105633; 1UG3HL146935-01A1 (NIH); 1U24HL146938-01A1 (NIH)
Record Dates: First submitted 2020-12-03; First posted 2020-12-09 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Cardiac Arrest
Keywords: cardiac arrest; cardiopulmonary resuscitation; telephone CPR; dispatch CPR; out-of-hospital cardiac arrest; defibrillation
MeSH Terms: conditions — Heart Arrest; Out-of-Hospital Cardiac Arrest | interventions — Cardiopulmonary Resuscitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Enhanced Standard of Care) (Experimental): Mass community CPR/AED training, optimize 911 medical dispatch, improve first responder performance
  Interventions: Other: Rapid cardiac arrest recognition that triggers immediate priority EMS/first responder dispatch by 911 operators; Other: Systematic bystander resuscitation instruction by 911 operators; Other: Comprehensive community training of lay people in CPR and AED use.; Other: Optimized first responder performance including earlier use of AEDs.
- Control (Standard of Care) (No Intervention): Usual care, continuing standard quality improvement effort

INTERVENTIONS:
Other: Rapid cardiac arrest recognition that triggers immediate priority EMS/first responder dispatch by 911 operators — EMS first responders will recognize cardiac arrest and respond immediately, increasing time to dispatch
  Arms: Intervention (Enhanced Standard of Care)
Other: Systematic bystander resuscitation instruction by 911 operators — 911 operators will be able to describe how to administer CPR over the phone.
  Arms: Intervention (Enhanced Standard of Care)
Other: Comprehensive community training of lay people in CPR and AED use. — Training of lay people regarding CPR and AED use.
  Arms: Intervention (Enhanced Standard of Care)
Other: Optimized first responder performance including earlier use of AEDs. — First responders will recognize where AEDs are located and use them appropriately
  Arms: Intervention (Enhanced Standard of Care)

SUMMARY:
RACE-CARS is a real-world cluster-randomized trial designed to evaluate a multifaceted community and health systems intervention aimed to improve outcomes of out-of-hospital cardiac arrest. RACE-CARS will enroll 50 counties in North Carolina that are estimated to have a total of approximately 20,000 patients with cardiac arrest over a 4-year intervention period. County "clusters" will be randomized in a 1:1 ratio to intervention versus usual care. The trial duration is 7 years, which includes a 6-month start-up (including recruitment and randomization) period, a 12-month intervention training phase, a 4-year intervention period, a 12-month follow-up for to assess quality of life in survivors of OHCA, and a 6-month close-out and data analysis period.

ELIGIBILITY:
Inclusion Criteria:

* OHCA of non-traumatic etiology
* Patients who are pulseless on arrival of a first responder; or patients who become pulseless in the presence of a first responder; OR patients who have a pulse on arrival of EMS, where a successful defibrillation was previously administered by a bystander or first responder.

Exclusion Criteria:

* Untreated cardiac arrests, including arrests in which resuscitation efforts are not initiated or are terminated immediately upon arrival of EMS because the patient is not a viable candidate for resuscitation due to:

  1. injuries incompatible with life,
  2. the presence of rigor mortis or lividity,
  3. signs of decomposition, or
  4. the presence of a valid DNR.
* Private EMS transport that did not involve 911 dispatch (example: interfacility transport between nursing home and hospital).
* Arrest of clear and obvious traumatic etiology
* Bystander suspected cardiac arrest, where ROSC was achieved without the need for defibrillation or first responder CPR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20000 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Survival with good neurologic outcomes as measured by a CPC score of 1 or 2 at discharge | up to 12months
  Cerebral Performance Category (CPC)

SECONDARY OUTCOMES:
Percent of patients who receive CPR from a bystander as measured by EMS report | Baseline
Rate of Defibrillation before paramedics arrive as measured by bystander interview | Baseline

OTHER OUTCOMES:
Percent of cardiac arrest patients whose cardiac arrests are recognized by 911-dispatcher through telephone call | Follow-up, up to 4 years
Percent of cardiac arrest patients with responders who receive CPR instructions by 911-dispatcher through telephone call | Follow-up, up to 4 years
Survival rate as measured by medical record abstraction | Follow-up, up to 4 years
Change in Neurologic disability as measured by Modified Rankin Score | 3 months, 12 months
  The Modified Rankin Score is a 6 point likert scale, with 0 being "No symptoms" and 6 being "Dead"
Change in Quality of life as measured by the SF-36 | 3 months, 12 months
  The SF-36 is Is a health-related quality-of-life questionnaire consisting of thirty six questions that measure eight health domains to assess physical and mental health. Physical health-related domains include General Health (GH), Physical Functioning (PF), Role Physical (RP), and Body Pain (BP).
Change in Quality of life as measured by the EQ-5D-5L | 3 months, 12 months
  The EQ-5D-5L is Quality of Life instrument measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Granger, MD, Principal Investigator — Duke University
Locations (1):
- Duke, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No